CLINICAL TRIAL: NCT06716541
Title: Biodegradable Stents Versus Plastic Stents for Treatment of Biliary Anastomotic Strictures in Liver Transplant RecipIents
Brief Title: Biodegradable Stents in Liver Transplant RecipIents for Treatment of Biliary Anastomotic Strictures
Acronym: BRILLIANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Tomas Hucl, Chairman, Department of Gastroenterology and Hepatology, Institute for Clinical and Experimental Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKEM BDS
Record Dates: First submitted 2024-11-25; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Liver Transplant, Complications; Biliary Anastomotic Stenosis; Endoscopic Retrograde Cholangiopancreatography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Management of anastomotic biliary strictures with biodegradable stents (Experimental): Initially, a single biodegradable stent is used for treatment of an anastomotic biliary stricture. If needed, this may be followed by usage of another biodegradable stent or plastic stents.
  Interventions: Procedure: ERCP implantation of a biodegradable stent; Procedure: ERCP implantation of plastic stents
- Management of anastomotic biliary strictures with multiple plastic stents in (Active Comparator): Multiple plastic stents are used for treatment of an anastomotic biliary stricture.
  Interventions: Procedure: ERCP implantation of plastic stents

INTERVENTIONS:
Procedure: ERCP implantation of a biodegradable stent — Endoscopic retrograde cholangiopancreatography (ERCP) with placement of a biodegradable stent to treat anastomotic biliary stricture (possibly combined with removal of previous plastic stents).
  Arms: Management of anastomotic biliary strictures with biodegradable stents
Procedure: ERCP implantation of plastic stents — Endoscopic retrograde cholangiopancreatography (ERCP) with placement of a plastic stent or multiple stents to treat anastomotic biliary stricture (possibly combined with removal of previous plastic stents).

SUMMARY:
Biliary complications after liver transplantation (LT) remain common and are associated with higher morbidity in liver transplant recipients and liver graft failure. Anastomotic biliary strictures are the most common biliary strictures after LT. Today, the gold standard for treatment remains endoscopic retrograde cholangiopancreatography (ERCP) with either multiple plastic stenting (MPS) or fully covered metal stents. These methods have disadvantages such as the need for repeated ERCP procedures, high costs or the risk of migration.

Biodegradable stents (BDS) are a novel type of stents made from various synthetic polymers or their copolymers, which are now being used in a variety of medical fields, including the pancreatobiliary tract.The use of biodegradable stents has shown good potential in the treatment of benign biliary strictures. However, overall data on their endoscopic use in liver transplant recipients, particularly in the treatment of anastomotic biliary strictures, are scarce. Most studies have either been in animal models, using percutaneously implanted stents, or in non-transplanted patients. There are no randomised controlled trials investigating their use in LT patients. Based on the available evidence, the use of BDS in the treatment of anastomotic biliary strictures in liver transplant recipients appears to be a promising technique that may be as effective as the standard treatment with MPS, but may reduce the number of ERCP procedures and eliminate the risk of migration.

The aim of this randomised prospective study is to compare the difference in rates of anastomotic stricture resolution between the active (BDS) and control (MPS) groups to demonstrate non-inferiority of the biodegradable stents. Outcomes will be classified as complete resolution (no significant stricture at the anastomotic site on imaging and resolution of cholestasis), significant response (relative stricture and resolution of cholestasis) or failure (persistent stricture and/or persistent cholestasis). Secondary outcomes are technical feasibility, immediate and late complications.

DETAILED DESCRIPTION:
Liver transplantation (LT) is nowadays a standard treatment method of end-stage liver disease, primary liver cancer and acute liver failure.

Biliary complications (BCs) following liver transplantation are the leading source of morbidity and liver graft failure and are associated with up to 10% mortality rate. The incidence of BCs remains high, being reported in 10-25% in cadaveric donors (DDLT) and in more than 30% in living donor liver transplantations (LDLT), despite improved both preoperative and postoperative care and enhanced surgical technique. Anastomotic biliary strictures (ABS) are together with bile leaks the most common biliary complication occurring any time after LT, but being primarily found within the first year LT. The incidence ranges between 5-15% in DDLT and 13-36% in LDLT. Anastomotic strictures are typically present at the site of anastomosis, tend to be short, single and constitute up to 86% of all biliary strictures. The clinical presentation can differ from patients being asymptomatic to some presenting with symptoms of biliary obstruction (jaundice, fever, chills, nausea, abdominal pain). The clinical picture can resemble also other conditions and it is important to differentiate biliary complication (BC) from other similarly presenting entities such as acute rejection, hepatic artery thrombosis, recurrence of primary sclerosing cholangitis or acute hepatitis). The gold standard for diagnosis of BCs is MRCP with reported sensitivity and specificity of up to 95%.

The first line therapy of BCs is endoscopic retrograde cholangiopancreatography (ERCP), in case of failure or altered anatomy percutaneous approach may be indicated. If both methods fail surgery is required. ERCP is an invasive endoscopic technique used primarily for therapy of pancreatobiliary tract. It is associated with risk of complications such as acute pancreatitis, bleeding, acute cholangitis or in rare cases perforation.

There are two standard approaches in the treatment of anastomotic biliary strictures, similarly to the treatment of other benign strictures of the bile duct. First, the use of multiple plastic stents (MPS) requiring their repeated endoscopic exchanges may be employed. Alternatively, a single self-expandable metal stent is placed for a longer period of time.

The endoscopic therapy of anastomotic strictures using multiple plastic stents typically requires multiple stent exchanges, starting with placing a single stent and adding multiple stents during further sessions. The sessions are scheduled every 1 to 3 months. The resolution of the anastomotic stricture is usually achieved in 12months, exposing the patient typically to 3-4 ERCP procedures. MPS technique was firstly described and put in practice in a single center study by Costamagna et al. with clinical success rate in 89%. After that many other studies have been published regarding this topic, including a meta-analysis, where the resolution rate of strictures were reported in 94%-100%. Finally in 2017 by Koksa et al. was reported a review demonstrating that in patients with more than 12 months of stenting, with higher total number of stents and number of stents inserted per session, a higher resolution rate and a lower recurrence rate were showed. Alternative option for the endoscopic treatment of ABS is the use of a single fully covered self-expandable metal stent (FC-SEMS), in studies showing similar rates of ABS resolution compared to MPS method with the advantage of not repeating ERCP to place multiple stents, although with higher risk of migration.

The use of endoscopically inserted biodegradable stents is a novel technique with a potential to overcome some downsides of standard treatment with MPS and FC-SEMS. Biodegradable stents are made of different synthetic polymers or their co-polymers. First use of biodegradable stents in the GI tract was described in the setting of an esophageal stricture in 1996 and was later used in small intestine and colon for benign strictures. In the pancreatobiliary tract biodegradable stents have begun to be used in the recent years, mostly for benign biliary strictures such as those caused by chronic pancreatitis and in postoperative cystic duct leaks. Most of the reported experience comes from percutaneously inserted stents. The experience with endoscopic insertion of biodegradable stents is very limited and the data about use of biodegradable stents in liver transplant recipients are extremely scarce.

A systematic review on the use of biodegradable stents in biliary tract by Siiki at al. reviewed studies from 1997 to 2017. This review included 12 animal and 7 human studies. In human studies biodegradable stents were inserted in 4 studies percutaneously and in 3 studies endoscopically. The main indications were benign biliary strictures, postoperative cystic duct leaks, leaks from hepaticojejunal anastomosis, strictures of hepaticojejunal anastomosis, bilioenteric anastomosis strictures or chronic pancreatitis. In all studies stents made out of polydioxanone with time of degradation between 3-6 months were used. The studies proved good feasibility and safety of BDS in both animal and human setting and demonstrated their successful use in the treatment of benign biliary strictures and cystic bile duct leaks. In the first and biggest study with the endoscopic use of biodegradable stents in humans in treatment of cystic duct leaks and benign biliary strictures (BBS), the overall clinical success rate in treatment of BBS was noted in 83% with no secondary hyperplastic strictures. Surprisingly quite high rate of acute cholangitis occurred, in 23% after 90 days, although all cases were mild.

In another recent systematic review and metanalysis by Almeida et al. biodegradable stents were compared to multiples plastic stent implantation in benign biliary strictures. In total 9 studies met the inclusion criteria and were analyzed. Biodegradable stent group (BDBS) consisted of one retrospective and two prospective cohort studies, where stents were deployed both endoscopically and percutaneously with a minimal follow up of 20,8 months. In contrast the MPS group consisted of one randomized control trial comparing the use of multiple plastic stents to FCSEMS for different types of benign biliary strictures, and 5 cohort studies from which were 4 retrospective and one was prospective with a minimal follow up of 78,4 months. The overall success rate to achieve long-term stricture resolution was 83% for the BDBS group and 84% for the MPS group. The average number of interventions in the MPS group was 3 in contrast to 1 in the BDBS group (per case). In a majority of cases the stents were placed percutaneously and only one cohort study included endoscopically released BDBS (13 patients). The treatment-related complication rate was reported for acute cholangitis, acute pancreatitis, stent migration and abdominal pain and was 24,1%, 0,7 %, 1,5 %, 0, 8% for BDBS and 6,1%, 2,7%, 6,8% and 6,8 % for MPS.

An observational single center study by Dopazo et al. reported 20 adult and pediatric patients where BDS were used for benign biliary strictures after liver transplantation using a transhepatic approach. The overall feasibility was 100%, the overall clinical success including both anastomotic and nonastomotic strictures was 75%. The clinical success was higher in anastomotic strictures (81,25%). Only one case of acute pancreatitis was observed.

Based on the available evidence, BDS have shown promising results with good stent patency, feasibility, efficacy and safety profile. Therefore, BDS may represent a novel treatment modality and an alternative to current techniques in the management of biliary anastomotic strictures with a reduced number of ERCPs. However, prospective comparative data are needed.

The investigators aim to compare the use of biodegradable stents with the multiple stenting technique using plastic stents for the treatment of biliary anastomotic strictures and to demonstrate the non-inferiority of biodegradable stents, as well as the safety profile and technical feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Liver transplant recipients
* Duct-to-duct biliary anastomosis
* Anastomotic biliary stricture (cholestasis unexplained by other causes and/or liver biopsy showing altered biliary drainage and/or anastomotic stricture on MRCP)
* Signed informed consent

Exclusion Criteria:

* Hepaticojejunoanastomosis
* Physical and/or psychological inability to understand the aims of the research and to adequately cooperate
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Persisting anastomotic stricture resolution | 12+6 months
  Rate of resolution of the anastomotic stricture as confirmed by Endoscopic retrograde cholangiopancreatography (ERCP) or Magnetic Resonance Cholangiopancreatography (MRCP) examination within 12 months since the initial procedure and persistence of the resolution (confirmed by MRCP) 6 months after the initial resolution.
  Resolution of anastomotic stricture is defined as all of the following simultaneously:
  * no need of further restenting
  * residual narrowing of lumen less than 20%)
  * alkaline phosphatase (ALP) below two times the upper limit of normal (unless a cause of the increase other than the anastomotic stricture is identified)
Number of ERCPs | 12 months
  The total number of ERCPs required for the stricture resolution

SECONDARY OUTCOMES:
Initial anastomotic stricture resolution | 12 months
  Rate of resolution of the anastomotic stricture as confirmed by Endoscopic retrograde cholangiopancreatography (ERCP) or Magnetic Resonance Cholangiopancreatography (MRCP) examination within 12 months since the initial procedure.
  Resolution of anastomotic stricture is defined as all of the following simultaneously:
  * no need of further restenting
  * residual narrowing of lumen less than 20%)
  * alkaline phosphatase (ALP) below two times the upper limit of normal (unless a cause of the increase other than the anastomotic stricture is identified)
Technical feasibility | 12 months
  Specific technical features related to the biodegradable stent (loadability, pushability, stent deployment, fluoroscopic visibility) and overall technical performance compared to commonly used plastic stents will be evaluated by endoscopists using a questionnaire at the end of the treatment period.
Safety | 12 months
  Device or procedure related adverse events (bleeding, perforation, cholangitis, pancreatitis, stent migration)
Number of stents placed | 12 months
  The total number of stents placed during ERCPs
Duration of stenting | 12 months
  The duration of the stenting period measured in months from the first to the last ERCP procedure.
Degradation of biodegradable stents | 6 months
  Absence of signal void in common bile duct at MRCP at 6 months in biodegradable stents group
Quality of life | 12 months
  Validated questionnaire investigating quality of live post intervention/s
Cost | 12 months
  Costs associated with the performed procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Hucl, Prof, Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (1):
- Institute for Clinical and Experimental Medicine, Department of Gastroenterology and Hepatology, Prague, Czechia